CLINICAL TRIAL: NCT05402566
Title: MRI Assessment of Impaired Glucose Metabolism in Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DMI-AD
Record Dates: First submitted 2022-05-25; First posted 2022-06-02 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2022-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healhy volunteers: Repeated MRI and DMI for simplification of protocols. Repeated within 6 +/- 2 weeks.
  Interventions: Diagnostic Test: Deuterium metabolic imaging
- Alzheimer's disease patients: MRI and DMI to assess cerebral glucose metabolism. Single examination. Compared with PET.
  Interventions: Diagnostic Test: Deuterium metabolic imaging
- Healthy controls: MRI and DMI for comparison with AD patients.
  Interventions: Diagnostic Test: Deuterium metabolic imaging

INTERVENTIONS:
Diagnostic Test: Deuterium metabolic imaging — MRI after oral administration of 75g of [6,6'-2H2]glucose.

SUMMARY:
Diseases of dementia are chronic, untreatable, and cause a massive burden of morbidity. In this proposal, we seek to tackle the problem of better, earlier, and more efficient diagnosis using deuterium metabolic imaging (DMI). The study is divided in two sub-studies: 1) optimization and simplification of DMI protocols, and 2) a cross-sectional study of DMI in Alzheimer's patients and healthy controls.

ELIGIBILITY:
Inclusion criteria:

AD-patients:

* Aged 55-85 years.
* Male or female.
* AD diagnosis by the NIA-AA 2011 research criteria.8
* Able to give written informed consent.
* Mini-mental state examination (MMSE) equal to or above 18.9
* Brain FDG-PET performed at Aarhus University Hospital consistent with AD.

Healthy participants:

* Aged 18-85 years.
* Male or female.

Exclusion criteria:

All participants:

* Diabetes or any other metabolic disease.
* Other significant brain disease:

  * Strokes.
  * Tumors.
  * Chronic small vessel disease (clinically suspected, or Fazekas ≥ 2 if clinical MRI is available).
  * Epilepsy.
  * Other neurodegenerative or -inflammatory disease.
* Contraindications for MRI:

  * Pacemaker, neurostimulator or cochlear implant.
  * Metal foreign bodies such as fragments and irremovable piercings.
  * Unsafe medical implants (safety of heart valves, hips and the like must be confirmed).
  * Claustrophobia.
  * Largest circumference including arms > 160 cm.
* Pregnant - women must be post-menopausal or confirmed non-pregnant by an onsite test.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In sub-study 1, the population is composed of healthy volunteers. In sub-study 2, patients with Alzheimer's disease and healthy age-matched controls are recruited.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Deuterium Metabolic Imaging | Up to 150 mins after 2H-glucose ingestion
  Glucose concentration in whole-brain referenced to baseline scan (sub-study 1).
Deuterium Metabolic Imaging | Up to 150 mins after 2H-glucose ingestion
  Lactate concentrations in whole-brain referenced to baseline scan (sub-study 1).
Deuterium Metabolic Imaging | Up to 150 mins after 2H-glucose ingestion
  Glx concentrations in whole-brain referenced to baseline scan (sub-study 1).
Deuterium Metabolic Imaging | Up to 150 mins after 2H-glucose ingestion
  Lactate/glx ratio in the tempo-parietal cortex (sub-study 2).
Deuterium Metabolic Imaging | Up to 150 mins after 2H-glucose ingestion
  Lactate/glx ratio in the hippocampus (sub-study 2).
Deuterium Metabolic Imaging | Up to 150 mins after 2H-glucose ingestion
  Lactate/glx ratio in the posterior cingulum (sub-study 2).

SECONDARY OUTCOMES:
Deuterium Metabolic Imaging | Up to 150 mins after 2H-glucose ingestion
  Simpler DMI quantifications, including reference to external phantoms and internal reference, in the same regions defined in primary outcomes.
Blood samples | Up to 150 mins after 2H-glucose ingestion
  Glucose
Blood samples | Up to 150 mins after 2H-glucose ingestion
  2H-enrichment
FDG-PET from the records (sub study 2) | At time of Deuterium Metabolic Imaging
  Brain glucose uptake
Cognitive tests from the records (sub study 2) | At time of Deuterium Metabolic Imaging
  The Mini-Mental State Exam (0-30, 30 is best)
Cognitive tests from the records (sub study 2) | At time of Deuterium Metabolic Imaging
  Addenbrooke's Cognitive Examination (0-100, 100 is best)
Cerebrospinal fluid biochemistry from the records (sub study 2) | At time of Deuterium Metabolic Imaging
  Total tau protein
Cerebrospinal fluid biochemistry from the records (sub study 2) | At time of Deuterium Metabolic Imaging
  Phosphorylated tau
Cerebrospinal fluid biochemistry from the records (sub study 2) | At time of Deuterium Metabolic Imaging
  Amyloid

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after study completion and full anonymization.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After study is completed.

REFERENCES:
- [Derived] Bogh N, Vaeggemose M, Schulte RF, Hansen ESS, Laustsen C. Repeatability of deuterium metabolic imaging of healthy volunteers at 3 T. Eur Radiol Exp. 2024 Mar 13;8(1):44. doi: 10.1186/s41747-024-00426-4. PMID 38472611